CLINICAL TRIAL: NCT03826004
Title: Effect of Histamine H1 Receptor Antagonist Clemastine in Cardiovascular Surgery With Cardiopulmonary Bypass: A Pilot Study
Brief Title: Clemastine in Cardiovascular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, SHI Jia, Assoticate Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Clemastine Pilot Study
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Efficacy and Safety
Keywords: Cardiovascular Surgery; Histamine H1 Receptor Antagonist; Anaphylaxis
MeSH Terms: conditions — Anaphylaxis | interventions — Clemastine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Saline solution 2ml before anesthetic induction
  Interventions: Drug: Saline Solution
- Clemastine (Experimental): Clemastine fumarate 2mg/2ml before anesthetic induction
  Interventions: Drug: Clemastine

INTERVENTIONS:
Drug: Clemastine — Clemastine fumarate 2mg/2ml intramuscular injection is administrated into the gluteus maximus muscle
  Arms: Clemastine
Drug: Saline Solution — Saline solution 2ml intramuscular injection is administrated into the gluteus maximus muscle
  Arms: Placebo

SUMMARY:
In this study, a prospective, randomized, double-blind pilot trial designed to evaluate the effect of histamine H1 receptor antagonist clemastine on perioperative anaphylaxis in cardiovascular surgery with cardiopulmonary bypass, especially for the efficacy and safety on reducing heparin and protamine associated anaphylaxis.

DETAILED DESCRIPTION:
In this study, a prospective, randomized, double-blind pilot trial designed to evaluate the effect of histamine H1 receptor antagonist clemastine on perioperative anaphylaxis in cardiovascular surgery with cardiopulmonary bypass, especially for the efficacy and safety on reducing heparin and protamine associated anaphylaxis.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* Receiving selective cardiovascular surgery with cardiopulmonary bypass due to coronary, valvular or congenital heart disease
* Written informed consent obtained.

Exclusion Criteria:

* Previous history of cardiac surgery
* Allergy to clemastine, antihistamines with similar chemical structure or any excipient (sorbitol, sodium citrate, propylene glycol, ethanol)
* Myasthenia gravis
* Porphyria patients
* Bronchial asthma
* Usage of monoamine oxidase (MAO) inhibitors
* Pregnant or lactating women
* Mentally or legally disabled patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Histamine concentration in plasma | Perioperative period
  Plasma histamine concentration evaluated by ELISA

SECONDARY OUTCOMES:
Blood pressure | Perioperative period
  Invasive blood pressure of radial artery: systolic, diastolic and mean pressure
Airway pressure | Perioperative period
  Airway pressure: peak and plat
Skin manifestation | Perioperative period
  Rate of skin manifestations, including wheal, papules, maculopapules, etc
Arrhythmia | Perioperative period
  Rate of perioperative arrhythmia, especially tachycardia
Specific symptoms | Perioperative period
  Rate of specific symptoms, including fatigue, sleepiness, dizziness, headache, stomach pain, constipation, nausea, dry mouth

CONTACTS AND LOCATIONS:
Overall Officials: Jia Shi, M.D., Study Chair — Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC
Locations (1):
- Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC, Beijing, Beijing Municipality, China